CLINICAL TRIAL: NCT07379632
Title: Treatment Effects of Vertical Holding Appliance in Comparison to Zachrisson Transpalatal Arch on Anterior Open Bite Correction During Mixed Dentition: A Randomized Controlled Trial
Brief Title: Treatment Effects of Vertical Holding Appliance in Comparison to Zachrisson Transpalatal Arch on Anterior Open Bite Correction
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Ola Alaa Yehia, Master student, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 3-3-4
Record Dates: First submitted 2026-01-23; First posted 2026-01-30 (Actual); Last update posted 2026-01-30 (Actual); Status verified 2026-01

CONDITIONS: Anterior Open Bite in Mixed Dentition

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- vertical holding appliance (Active Comparator): a transpalatal arch with acrylic button
  Interventions: Device: Vertical holding appliance
- Zachrisson transpalatal arch (Experimental): a transpalatal arch with 2 posterior loops and 1 anterior loop
  Interventions: Device: Zachrisson transpalatal arch

INTERVENTIONS:
Device: Zachrisson transpalatal arch — transpalatal arch with 2 posterior loops and 1 anterior loop
  Arms: Zachrisson transpalatal arch
Device: Vertical holding appliance — transpalatal arch with arcylic button
  Arms: vertical holding appliance

SUMMARY:
The aim of the study is to assess the treatment effects of ZTPA versus VHA in the correction of anterior open bite in mixed dentition.

ELIGIBILITY:
Inclusion Criteria:

1. Children with the age rage from 6-12 years old.
2. Both male and female.
3. Class I and II skeletal and dental.
4. Skeletal anterior open bite.
5. Maxillary and mandibular incisors and upper first molars erupted.
6. Good oral hygiene.

Exclusion Criteria:

1. Systemic disease.
2. Missing teeth.
3. Previous orthodontic treatment.
4. Presence of posterior crossbites.

Ages: 6 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 38 (Estimated)
Dates: Start 2024-01-01 (Actual); Primary Completion 2025-06-01 (Actual); Study Completion 2026-06-01 (Estimated)

PRIMARY OUTCOMES:
Vertical skeletal measurements using cephalometric analysis | 9 months

SECONDARY OUTCOMES:
Overbite reduction | 9 months

CONTACTS AND LOCATIONS:
Overall Officials: ola a yehia, master student, Principal Investigator — Cairo University
Locations (1):
- Faculty of Dentistry Cairo University, Cairo, Egypt